CLINICAL TRIAL: NCT02966691
Title: Evaluation of Diagnostic Performance of VisioCyt® Test, in Case of Suspicion of Urothelial Bladder Tumors
Acronym: VISIOCYT 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitadx (Other)
Collaborators: FONDATION FORCE POUR L'INNOVATION ET LA RECHERCHE EN SANTE (Unknown); SATT Paris Saclay (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00623-48
Record Dates: First submitted 2016-10-28; First posted 2016-11-17 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients 'sick' (Active Comparator): The patients of this arm have a clinical signs of bladder cancer with :
  * a positive result of bladder endoscopy
  * or an negative endoscopy and a positive result of the conventional cytology
  The intervention consists to collect an additional urine sample (50 ml), the day of the bladder endoscopy, which is performed during the current practice .This urine sample will be used for the preparation of cytology slides according to the Visiocyt protocol, in order to be digitized
  Interventions: Other: VisioCyt® diagnostic test
- Patients 'healthy' (Active Comparator): The patients of this arm have no suspicion of bladder cancer with negative results of their bladder endoscopy and conventional cytology.
  The intervention consists to collect an additional urine sample (50 ml), the day of the bladder endoscopy, which is performed during the current practice . This urine sample will be used for the preparation of cytology slides according to the Visiocyt protocol, in order to be digitized.
  Interventions: Other: VisioCyt® diagnostic test
- Patients 'monitoring' (Active Comparator): The patients of this arm have a history of bladder cancer, but the results of their follow up examinations (cytologic and endoscopic) are negative (no tumor).
  The intervention consists to collect an additional urine sample (50 ml), the day of the bladder endoscopy, which is performed during the current practice . This urine sample will be used for the preparation of cytology slides according to the Visiocyt protocol, in order to be digitized.
  Interventions: Other: VisioCyt® diagnostic test

INTERVENTIONS:
Other: VisioCyt® diagnostic test — The cytology slides obtained from the current practice will be compared to the slides obtained with the Visiocyt protocol, for each arm.

SUMMARY:
This clinical study is designed to evaluate the diagnostic performance of VisioCyt test, which would improve the early diagnosis of bladder cancer in order to optimize the management of individual patients as part of a cancer diagnostic monitoring. The diagnostic method of VisioCyt® device is based on the analysis by transmission and fluorescence, of urinary cytology slides prepared according to the protocol VisioCyt.

DETAILED DESCRIPTION:
This clinical trial is divided into two main phases:

I. The first one involves the construction of better image processing algorithm from a learning sample. The learning sample will include 600 virtual slides made from the urine sample of the first 600 patients enrolled.

II. The second one, will evaluate from an evaluation sample, the diagnostic performance of the test VisioCyt, to identify patients with versus without bladder tumors, using as comparator the results of the examination of reference: histology. The evaluation sample will include 400 slides, made from the urine sample of the last 400 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient affiliated to a social security system
* Patient able to understand the protocol.
* Signature of patient consent form before the start of the study
* Negative urine culture
* Patient for which is programmed a bladder Endoscopy for :

  * suspected bladder cancer (de novo, monitoring or relapse)
  * Exploration lower urinary tract excluding a suspected bladder cancer or prostate cancer

Exclusion Criteria:

* Age <18 years
* Ongoing Urinary tract infection untreated
* Private person of liberty or under guardianship (including guardianship)
* Bladder cancer excluding urothelial carcinoma
* Carcinoma of high urinary tract, associated
* Lithiasis pathology
* Patient who underwent renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1360 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Identification and classification of cells with the VisioCyt test to create an image processing algorithm | 9 months
  * Identification and classification of cells, taking the Paris System in 2016 as a referential
Identification of presence or absence of a membrane fluorescence perished with the VisioCyt test to create an image processing algorithm | 9 months
  presence or absence of a membrane fluorescence perished, on slides
sensitivity of urinalysis by VisioCyt test | through the study completion
  number of patients "declared positive" with the VisioCyt test among the patients actually suffering from bladder carcinoma
specificity of urinalysis by VisioCyt test | through the study completion
  number of patients "declared negative" with the VisioCyt test among the really healthy patients

SECONDARY OUTCOMES:
sensitivity of urinalysis by VisioCyt test according to the cell grade of the patients | through the study completion
  number of patients "declared positive" with the VisioCyt test among the patients with a "low grade" or "high grade" bladder carcinoma
sensitivity of urinalysis by VisioCyt test according to medical history of the patients | through the study completion
  number of patients "declared positive" with the VisioCyt test among the patients with a first diagnosis of bladder carcinoma or among patients with a previous bladder carcinoma under monitoring
comparison of the sensitivity of the urinalysis by VisioCyt test versus conventional urine cytology | through the study completion
  number of patients "declared positive" with the VisioCyt test versus patients "declared positive" with the conventional urine cytology
comparison of the specificity urinalysis by VisioCyt test versus conventional urine cytology | through the study completion
  number of patients "declared negative" with the VisioCyt test versus patients "declared negative" with the conventional urine cytology

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Hôpital d'Antony, Antony
  - Clinique " la Châtaigneraie ", Beaumont
  - CHU de Besançon, Besançon
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Clinique BeauSoleil, Montpellier
  - Hôtel Dieu, CHR de Nantes, Nantes
  - CHU Caremeau, Nimes, Nîmes
  - Hôpital Cochin, Paris
  - CHU Rennes, Rennes
  - Hôpital Foch, Suresnes
  - Hopital Rangueil, Toulouse
  - CHRU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No